CLINICAL TRIAL: NCT05737498
Title: Efficacy of Transcranial Direct Current Stimulation (tDCS) on Working Memory in College Going Students
Brief Title: Transcranial Direct Current Stimulation (tDCS) on Working Memory in College Going Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Subhasish Chatterjee, Assistant Professor ( Department of physiotherapy), Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IEC-2322
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Working Memory Deficits
Keywords: working memory, immediate memory
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Transcranial direct current stimulation will use to deliver a constant direct current through two surface electrodes, Anodal stimulation will applied according to the 10-20 international system for EEG electrode placement, over F3 of the dorsolateral prefrontal cortex (DLPFC), while the cathode will placed over the contralateral supraorbital area with 1.5 ma intensity for 20 min with working memory task on alternate days for two weeks.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- memory task training group (No Intervention): working memory task training for 20 min for two weeks

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation will use to deliver a constant direct current through two surface electrodes, Anodal stimulation was applied according to the 10-20 international system for EEG electrode placement, over F3 of the dorsolateral prefrontal cortex (DLPFC), while the cathode was placed over the contralateral supraorbital area for 20 min, on alternate days for 2 weeks 6 sessions with working memory training task. the anode (positive) and the cathode (negative). To reduce resistance and minimize discomfort during application (the electrodes were covered in 35 cm2, saline-soaked sponges
  Other Names: working memory training task
  Arms: experimental

SUMMARY:
Working memory deficiencies, might make it difficult for students to recall instructions, complete complex activities, and grasp and follow directions solving a math problem or writing a sentence. The functions of working memory are critical for effective human activity. Transcranial direct current stimulation (tDCS) has grown in popularity and academic interest in recent years as a way to improve cognitive abilities. so there is need to determine the effect of tdcs on working memory in college going students.

ELIGIBILITY:
Inclusion Criteria:

1. College going students
2. Both male and female
3. Able to follow verbal commands

Exclusion Criteria:

1. Chronic skin problems.
2. Seizure and any neurological disorder
3. Any recent trauma or surgery
4. Any cardiovascular or pulmonary disease
5. Psychosomatic disorders

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Trail making test | changes between baseline to 2 weeks
  As the participant proceeds in an increasing sequence, he or she must alternate between numbers and letters. Subjects are challenged to link numbers and alphabets as quickly as possible. The examiner calls out errors as they happen so that the subject can finish the test without making any mistakes
Digit span test | changes between baseline to 2 weeks
  Digit Span Forward requires the child to repeat numbers in the same order as read aloud by the examiner, and Digit Span Backward requires the child to repeat the numbers in the reverse order of that presented by the examiner.